CLINICAL TRIAL: NCT04161638
Title: Weight Stigma in Women Who Are Obese: Assessing How an Acute Exposure to Stigma Negatively Impacts Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Linda Pescatello, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: H16-292HHC
Record Dates: First submitted 2019-11-06; First posted 2019-11-13 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Stigma, Social; Obesity; Cardiovascular Disease Risk Factor; Blood Pressure
MeSH Terms: conditions — Social Stigma; Obesity

STUDY DESIGN:
Intervention Model Description: Participants were randomized using www.randomization.com to either STIGMA at Visit 2 and NEUTRAL at Visit 3, or NEUTRAL at Visit 2 and STIGMA at Visit 3.
Who Masked: Participant
Masking Description: Due to the nature of the experimental manipulation in this study and to maintain validity, mild deception was necessary. Participants were told that the study was examining BP, HR, mood, and behavioral responses to various forms of media and were not informed specifically of the purpose until after they completed the study. In order to verify that the participants were unaware that their cardiovascular reactivity to a weight stigma exposure was being measured, a manipulation check was implemented wherein participants were asked to report what they believed the study purpose to be. No participants reported the true purpose of the study during the manipulation check. At the conclusion of the study, participants were debriefed about the true purpose of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Blood Pressure (Experimental): Ambulatory BP measurement was used to confirm the laboratory BP group classification according to the European Society of Hypertension. Participants were placed in the high blood pressure (HBP) group if they met any of the following criteria: 1) 19-hour average systolic BP/diastolic BP (SBP/DBP) > 130/80 mmHg, 2) daytime (awake) average SBP/DBP > 135/85 mmHg, or 3) nighttime (sleep) average SBP/DBP > 120/70 mmHg.
  Interventions: Behavioral: Stigma Video Exposure; Behavioral: Neutral video exposure
- Normal Blood Pressure (Experimental): Participants were placed in the normal BP (NBP) group if they met all of the following criteria: 1) 19-hour average SBP/DBP < 130/80 mmHg, 2) daytime (awake) average SBP/DBP < 135/85 mmHg, and 3) night-time (asleep) average SBP/DBP <120/70 mmHg.
  Interventions: Behavioral: Stigma Video Exposure; Behavioral: Neutral video exposure

INTERVENTIONS:
Behavioral: Stigma Video Exposure — The participants watched a 10 minute video on a computer screen that consisted of brief clips from popular television shows that depicted women with overweight and obesity and evoked negative weight-based stereotypes (e.g., clumsy, loud, and lazy). Both the high blood pressure and normal blood pressure arms participated in this intervention.
  Other Names: STIGMA
Behavioral: Neutral video exposure — The participants watched a 10 minute video on a computer screen that consisted of a series of clips depicting neutral scenes (e.g., insurance commercials). Both the high blood pressure and normal blood pressure arms participated in this intervention.
  Other Names: NEUTRAL

SUMMARY:
The current study examined the influence of an acute weight stigma exposure on cardiovascular reactivity among women with obesity and high blood pressure and women with obesity and normal blood pressure.

DETAILED DESCRIPTION:
The current study examined the influence of two video exposures, one containing scenes of weight stigma (STIGMA) and the other non-stigmatizing neutral (NEUTRAL) scenes, on cardiovascular reactivity as assessed by resting BP and ambulatory blood pressure (ABP) and heart rate (HR), among women with obesity and high BP (HBP) or normal BP (NBP). The investigators hypothesized that as a result of STIGMA compared to NEUTRAL, cardiovascular reactivity would be significantly greater immediately upon watching the video and persist outside of the laboratory over ambulatory conditions in women with obesity and HBP compared to women with obesity and NBP.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* BMI > 30 kg/m2
* No other known chronic cardiovascular or metabolic diseases besides hypertension

Exclusion Criteria:

* Pregnant or planned on becoming pregnant
* Took medications that may have affected the primary outcome of BP (e.g., stimulants for attention deficit hyperactivity disorder or steroids for asthma)
* Currently using tobacco products
* Diagnosed with an eating disorder

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Ambulatory systolic BP (SABP) reactivity | 19 hours (10 hours awake, 9 hours sleep)
  Ambulatory SABP reactivity was calculated as the change in hourly SABP values (mmHg) over the awake (10 hours), sleep (9 hours), and 19 hours minus average baseline SABP following STIGMA and NEUTRAL.

SECONDARY OUTCOMES:
Laboratory systolic blood pressure (SBP) reactivity | 20 minutes (2 minute intervals) before the exposure video; 10 minutes during the exposure video (2 min intervals); and 20 minutes following the exposure video (2 min. intervals).
  Laboratory SBP reactivity was calculated as the change in SBP in millimeters of mercury (mmHg) during the stigma video exposure (STIGMA) and the neutral video exposure (NEUTRAL) and 20-minute post-STIGMA and NEUTRAL minus baseline SBP.
Ambulatory diastolic BP (DABP) reactivity | 19 hours (10 hours awake, 9 hours sleep)
  Ambulatory DABP reactivity was calculated as the change in hourly DABP values (mmHg) over the awake (10 hours), sleep (9 hours), and 19 hours minus average baseline DABP following STIGMA and NEUTRAL.
Laboratory diastolic blood pressure (DBP) reactivity | 20 minutes (2 minute intervals) before the exposure video; 10 minutes during the exposure video (2 min intervals); and 20 minutes following the exposure video (2 min. intervals).
  Laboratory DBP reactivity was calculated as the change in DBP in millimeters of mercury (mmHg) during the stigma video exposure (STIGMA) and the neutral video exposure (NEUTRAL) and 20-minute post-STIGMA and NEUTRAL minus baseline DBP.
Laboratory heart rate (HR) reactivity | 20 minutes (2 minute intervals) before the exposure video; 10 minutes during the exposure video (2 min intervals); and 20 minutes following the exposure video (2 min. intervals).
  Laboratory HR reactivity was calculated as the change in HR in beats per minute (bpm) during the stigma video exposure (STIGMA) and the neutral video exposure (NEUTRAL) and 20-minute post-STIGMA and NEUTRAL minus baseline BP.
Ambulatory heart rate (HR) reactivity | 19 hours (10 hours awake, 9 hours sleep)
  Ambulatory heart rate (HR) reactivity was calculated as the change in hourly HR values (bpm) over the awake (10 hours), sleep (9 hours), and 19 hours minus average baseline HR following STIGMA and NEUTRAL.
Ambulatory rate pressure product (RPP) reactivity | 19 hours (10 hours awake, 9 hours sleep)
  Ambulatory RPP reactivity in mmHg*bpm was calculated as ambulatory SBP cardiovascular reactivity (mmHg) multiplied by ambulatory HR reactivity (bpm) (i.e., SBP x HR).
Laboratory rate pressure product (RPP) reactivity | 20 minutes (2 minute intervals) before the exposure video; 10 minutes during the exposure video (2 min intervals); and 20 minutes following the exposure video (2 min. intervals).
  Laboratory RPP reactivity in mmHg*bpm was calculated as laboratory SBP cardiovascular reactivity (mmHg) multiplied by laboratory HR reactivity (bpm) (i.e., SBP x HR).

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Taylor, PhD, Principal Investigator — University of Connecticut; Linda S Pescatello, PhD, Principal Investigator — University of Connecticut; Rebecca Puhl, PhD, Principal Investigator — University of Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Panza GA, Puhl RM, Taylor BA, Cilhoroz B, Himmelstein MS, Fernandez AB, Pescatello LS. The effects of an acute weight stigma exposure on cardiovascular reactivity among women with obesity and hypertension: A randomized trial. J Psychosom Res. 2023 Feb;165:111124. doi: 10.1016/j.jpsychores.2022.111124. Epub 2022 Dec 21. PMID 36571973